CLINICAL TRIAL: NCT03695783
Title: Impact of a Web-Based Decision Aid on Shared Decision-Making in Patients With Inflammatory Bowel Disease: The IBD&me Randomized Controlled Trial
Brief Title: The IBD&me Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Brennan Spiegel, Director, Health Services Research, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 37998665
Record Dates: First submitted 2018-09-26; First posted 2018-10-04 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Masking Description: Given the study design and intervention, it is not possible to ensure the blinding of patients and physicians. However, we will attempt to address the limitations resulting from a lack of blinding:
  * Patients and the physicians will be informed of the study protocol, but will not be provided accurate information about the specific primary outcome (i.e. comparison between IBD&me and the Crohn's & Colitis Foundation of America (CCFA) resource). The informed consent document will keep participants blind to the study goals.
  * Physicians will be kept blinded of the patient's assignment group until the clinic visit.
  * Data will be collected by an independent researcher. Study investigators and the data analyst will remain blinded until all follow-up data is obtained and the primary analysis is finalized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online decision aid called IBD&me (Experimental): IBD&me is an online, freely available tool that allows patients to explore decision-making around biologic therapies for IBD at their own pace. It includes an educational component and an interactive exercise with a series of ratings tasks that generates a personalized preferences report for patients to share and discuss with their physician.
  Interventions: Other: Online decision aid called IBD&me
- Standardized educational material (Active Comparator): PDF file corresponding to the CCFA's online resource on biologic therapies, which is a well-researched and clearly presented overview of IBD biologic therapies, but without an active shared-decision making component.
  Interventions: Other: Standardized educational material

INTERVENTIONS:
Other: Online decision aid called IBD&me — Patients randomized to IBD&me will be directed to go through the website at least 2 days before their clinic appointment, and will be asked to bring their personalized report with them to their upcoming visit.
  Arms: Online decision aid called IBD&me
Other: Standardized educational material — Patients randomized to the control arm will be sent a PDF file corresponding to the CCFA's online resource at least 2 days before their clinic appointment, and will be asked to bring it with them to their upcoming visit.
  Arms: Standardized educational material

SUMMARY:
Navigating the risk-benefit profiles of the various biologic options approved for inflammatory bowel disease (IBD) can be challenging for patients who are considering biologic therapies as a treatment option. Thus, there is a need for simple and efficient tools that elicit individual preferences and support the patient-provider interaction.

The principal objective of this study is to assess the impact of an online decision aid called IBD&me on patient perceptions of shared-decision making as compared to a standardized education arm.

DETAILED DESCRIPTION:
Context: Navigating the risk-benefit profiles of the various biologic options approved for inflammatory bowel disease (IBD) can be challenging for patients who are considering biologic therapies as a treatment option. Thus, there is a need for simple and efficient tools that elicit individual preferences and support the patient-provider interaction.

Objective: The principal objective of this study is to assess the impact of an online decision aid called IBD&me on patient perceptions of shared-decision making as compared to a standardized education arm.

Hypothesis: IBD&me, through optimizing shared-decision making (SDM) and improving the patient-provider interaction, will provide incremental benefits beyond those provided by high-quality educational material without an SDM tool.

Design: Pragmatic multicenter randomized controlled trial in IBD outpatient care

1. Intervention: IBD&me is an online, freely available tool that allows patients to explore decision-making around biologic therapies for IBD at their own pace
2. Control arm: Standardized, high-quality educational material from the Crohn's & Colitis Foundation

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have ulcerative colitis (UC), Crohn's disease (CD), indeterminate colitis, or inflammatory bowel disease unclassified (IBD-U)
* Have experienced IBD related symptoms in the 30 days before screening
* Considering discussing biologic therapies for controlling his or her IBD at the next clinic visit
* Have an IBD-related visit scheduled at least 7 days and no later than 3 months following screening

Exclusion Criteria:

* Does not speak English
* Does not have access to the Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2021-03-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Patient perceptions of shared decision-making | one day after the clinic visit
  To assess the impact of the IBD&me decision aid on patient perceptions of shared decision-making, compared to a standardized education arm. Patient perception of shared decision-making, as measured by the 9-item Shared Decision-Making Questionnaire (SDM-Q-9)

SECONDARY OUTCOMES:
Patient perceptions of decisional conflict | one day after the clinic visit
  Patient perceptions of decisional conflict, as measured using the informed and values clarity subscales of the Decisional Conflict Scale
Patient satisfaction | one day after the clinic visit
  Patient satisfaction as measured by four domains of the Patient Satisfaction Questionnaire relating to communication, general satisfaction, interpersonal manner, and time spent with the doctor (PSQ-18)
Disease control and IBD-related quality of life | at baseline and two months after the clinic visit
  Disease control and IBD-related quality of life, as measured by the IBD-Control questionnaire
Initiation or switch of a treatment | at baseline and two months after the clinic visit
  Questionnaire about IBD therapy use

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Spiegel, MD, MSHS, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No